CLINICAL TRIAL: NCT01577472
Title: Prospective Randomized Phase IV Study Comparing the Effect of Adding Clomiphencitrate Versus Placebo to a High Dose Versus a Minimal Dose GnRH Antagonist Protocol on the Number of Oocytes Collected From Women That Are Poor Responders
Brief Title: Efficacy Study Comparing the Effect of Clomiphencitrate to an Antagonist Protocol
Acronym: CANTAPOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CANTAPOR_2012
Record Dates: First submitted 2012-04-05; First posted 2012-04-13 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Female Infertility; Ovarian Insufficiency
Keywords: female infertility; poor ovarian response; controlled ovarian hyperstimulation; IVF; Antagonist protocol
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- High Dose Clomiphencitrat (Active Comparator): 450 IU Merional® plus 100mg Serophene®
  Interventions: Drug: High Dose Clomiphencitrat
- Low Dose Clomiphencitrat (Active Comparator): 150 IU Merional® plus 100mg Serophene®
  Interventions: Drug: Low Dose Clomiphencitrat
- High Dose Placebo (Placebo Comparator): 450 IU Merional® plus Placebo
  Interventions: Drug: High Dose Placebo
- Low Dose Placebo (Placebo Comparator): 150 IU Merional® plus Placebo
  Interventions: Drug: Low dose Placebo

INTERVENTIONS:
Drug: High Dose Clomiphencitrat — 100mg of clomiphencitrate(Serophene®) are added to a high dose of HMG (450 IU of Merional®) in the early follicular phase of the stimulation (day 3 to 7).
  Arms: High Dose Clomiphencitrat
Drug: Low Dose Clomiphencitrat — 100mg of clomiphencitrate(Serophene®) are added to a low dose of HMG (150 IU of Merional®) in the early follicular phase of the stimulation (day 3 to 7).
  Arms: Low Dose Clomiphencitrat
Drug: High Dose Placebo — Placebo is added to a high dose of HMG (450 IU of Merional®) in the early follicular phase of the stimulation (day 3 to 7).
  Arms: High Dose Placebo
Drug: Low dose Placebo — Placebo is added to a low dose of HMG (150 IU of Merional®) in the early follicular phase of the stimulation (day 3 to 7).
  Arms: Low Dose Placebo

SUMMARY:
The aim of this study is to assess the oocyte yield of infertile women with suspected or known poor ovarian reserve (POR) undergoing a GnRH antagonist protocol for IVF with Merional® starting either with a low (150 IU) or a high dose (450 IU) and adding 100mg of CC (Serophene®) in the early follicular phase of the stimulation (day 3 to 7). To date no RCT has been conducted to compare the reproductive outcome of patients with POR as defined by the ESHRE Bologna criteria after controlled ovarian hyperstimulation with HMG in an GnRH antagonist protocol using low doses versus high doses of HMG and adding CC versus placebo. We hypothesize that adding 100 mg of CC on day 3-7 to a HMG antagonist protocol will lead to an additional increment of endogenous GT thus increasing the oocytes yield after controlled ovarian stimulation due to higher endogenous gonadotropin secretion.

ELIGIBILITY:
Inclusion Criteria:

* Age: >18 years < 43 years
* BMI: ≥ 18 ≤ 32 kg/m2
* Poor responder as defined by ESHRE working group

Exclusion Criteria:

* Age < 18 und > 43 years
* Pregnancy
* Breast feeding
* Uterine conditions interfering with endometrial proliferation and embryo implantation (submucous fibroids or polyps)
* Women diagnosed with PCOS according to the Rotterdam criteria
* Hyperprolactinaemia - untreated
* Both ovaries not accessible transvaginally for oocyte pick up
* Ovarian cysts of unclear dignity
* Evidence of hydrosalpinx on ultrasound
* Clinically significant severe systemic disease that are incompatible with pregnancy
* Known or suspected hypersensitivity to the active substances (gonadotrophins, ganirelix, progesterone, clomiphencitrate)
* Untreated thyroid or adrenal disorders
* Bleeding disorders
* Cancer
* Severe renal or hepatic dysfunction
* Necessity to take medication that could influence ovarian stimulation
* History of OHSS in prior IVF cycle

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
number of collected oocytes | 1 year

SECONDARY OUTCOMES:
Implantation rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca E Moffat, MD, Principal Investigator — University Hospital Basel, Women's Clinic
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Moffat R, Hansali C, Schoetzau A, Ahler A, Gobrecht U, Beutler S, Raggi A, Sartorius G, De Geyter C. Randomised controlled trial on the effect of clomiphene citrate and gonadotropin dose on ovarian response markers and IVF outcomes in poor responders. Hum Reprod. 2021 Mar 18;36(4):987-997. doi: 10.1093/humrep/deaa336. PMID 33367742